CLINICAL TRIAL: NCT03435263
Title: Hospital Admission Versus Home Management in Women Premature Rupture of Membranes:RCT
Brief Title: Hospital Admission Versus Home Management in Women With Premature Rupture of Membranes :RCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, ahmed mahmoud hussein, lecturer of obstetrics and gyncology. MD, Ain Shams University
Other Study IDs: ain shams university protocol
Record Dates: First submitted 2018-02-06; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Management of Women With PROM at Term
Keywords: premature rupture of membranes
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hospital admission group B: Women presented with premature rupture of membranes will be admitted at hospital.
- home management group A: home management
  Interventions: Other: home management

INTERVENTIONS:
Other: home management — pregnant women presented with PROM will be randomized into 2 groups group a will be discharged home after initial assessment and group B will be admitted to hospital as usual
  Groups: home management group A

SUMMARY:
According to high tendency for admission of cases of premature rupture of membranes (PROM) for fear of maternal & fetal complications, we compare here between cases managed at hospital with other managed at home for if there any difference between in maternal and neonatal outcome.

DETAILED DESCRIPTION:
Premature rupture of membranes (PROM) refers to rupture of fetal membranes prior to onset of labor at term (> 37 weeks) (American college of obstetrician & gynecologist, 2007; Caughey et al., 2008).

A premature rupture of membranes (PROM) is observed in 8% of all pregnancies after 37 wk of gestational age,3% before and 5% after 37 weeks of gestation (Popowski et al., 2011;Keith, 2005) These membranes form an adjustable container for a developing and moving fetus, but it has limited life time, existing only to the point of programmed rupture at term, which is a normal event during the first stage of labor (Goldenberg and Rouse, 1998). As fetal membranes act as a barrier to ascending infection, so once membranes rupture both mother & fetus are at risk of infection and other complications (American college of obstetrician & gynecologist , 2007).

The latent period of labor is the time from rupture of membranes to the onset of effective uterine contractions, as this period tends to increase the risk of maternal and fetal infection, maternal infection termed chorioamnionitis which occurs in 3-5% of cases of PROM. While fetal infection occurs in about 15-20% in those with chorioamnionitis. Fetal infection may occur as septicemia, pneumonia, UTI, local infection as omphalitis (infection of the umbilical cord or conjunctivitis (Benedetto et al.,2004).

Other complications that may associated with PROM include umbilical cord prolapse in about 1.5% of cases of PROM. Placental abruption, caesarean delivery, postpartum hemorrhage and postpartum infection (Modena et al.,2004).

Correct diagnosis of PROM has great importance because failure to diagnose can lead to unwanted obstetric complications as chorioamnionitis, preterm birth. On the other hand over diagnose can lead to unnecessary intervention like hospitalization. The approach to diagnose rupture of membrane is clinical , with over 90% of cases being confirmed bases on the presence of suspicious history or ultrasonographic finding followed be documentation of fluid passing from the cervix (Hasan and Cevder et al., 2007).

The causes of PROM is not clearly understood, but the following risk factors that have been shown to increase the chance of its happening. In many cases, however no risk factors can be idintified.

1. Infection: UTI, STD, lower genital infection (ex: bacterial vaginosis).
2. Intrauterine infection.
3. Multiple previous pregnancies.
4. Cervical incompetency.
5. Hydramnios: too much AF.
6. Nutritional deficits.
7. Family history of PROM .(Ashley et al., 2003) . 8- Low socioeconomic status.

9-Multiple gestation: being pregnant with two or more fetuses at one time. 10- Previous preterm delivery. (Andrew et al.,2000) 11- Having had episodes of bleeding anytime during pregnancy. 12- Invasive procedure(ex: amniocentesis). 13- Being underweight. 14- Cigarette smoking during pregnancy(Jones., 2004) 15- Illicit drug use during pregnancy. 16- Having had PROM or preterm labor in previous pregnancy.(Parry., 2004) We observe in over 60% of the cases spontaneous labor begins within 24 hours, in 95% within 72 hours. often labor is induced after 24 hours because of the risk of maternal & neonatal is rising.

Majority of clinicians advise hospital care to allow monitoring and detection of problems. But for low risk patients fulfilling strict criteria sometimes home management is possible.

The initial management of a woman presenting with suspecting PROM should focus on confirming the diagnosis, validating the gestational age as maternal and fetal risks vary with the gestational age at time of membranes rupture as proved by (Morales and Talley. ,1993 ) .

It is important to make a distinction between term PROM and preterm PROM (PPROM) which is rupture of membranes before term (<37 weeks), as the conditions have different etiologies, risks and recommended management plans (Jones., 2004)

ELIGIBILITY:
Inclusion Criteria:

- Maternal age 20-35 years old. Singleton pregnancy. Patient presented with PROM. Gestational age >37 weeks. Estimated fetal weight 2.5-4 kg . Cephalic presentation. No evidence of chorioamnionitis. Reassuring tests of fetal wellbeing: non stress tests (CTG). No signs of infection: fever or tachycardia . Clear AF. No contraction.

Exclusion Criteria:

Maternal age < 20 or > 35 years old. Multiple pregnancy. Rupture of membranes before 37 weeks of gestation or postdate. Suspected IUGR. SuspectedFetal weight > 4 kg (suspected by clinical examination or ultrasound).

Congenital fetal anomalies. Malpresentation or malposition. Placental abnormalities. High risk pregnancy as hypertension, DM and pre-eclampsia . Evidence suggesting onset of spontaneous delivery (e.g.: vaginal bleeding or uterine contractions).

Previous cesarean section or other uterine surgery. Presence of signs of chorioamnionitis. Presence of signs of fetal distress. Meconium stained liquor. Mental condition rendering

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women at term pregnancy with PROM
Study Population: This study will be carried out on 72 pregnant women recruited from Obstetric Department of Ain Shams University Maternity Hospital presented with PROM after 37 weeks of gestation
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
latency period. | up to 24 hours
  time form rupture of membranes till starting labor

SECONDARY OUTCOMES:
NICU admission | first 24 hours after delivery
  neonatal ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: ahmed mahmoud hussein, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No